CLINICAL TRIAL: NCT05473728
Title: A Nationwide Multi-center Epidemiology Study and Risk Factor Analysis on Chronic Post-surgical Pain After Video-assisted Thoracic Surgery
Brief Title: Epidemiology Study and Risk Factor Analysis on Chronic Post-surgical Pain After Video-assisted Thoracic Surgery
Status: Completed | Type: Observational
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other); Tianjin Medical University Cancer Institute and Hospital (Other); First Affiliated Hospital of Chongqing Medical University (Other); Xiangya Hospital of Central South University (Other); Shanghai Chest Hospital (Other); The Affiliated Hospital of Inner Mongolia Medical University (Other); The people's hospital of Xinjiang (Unknown); Cancer hospital affiliated to Xinjiang Medical Universtity (Unknown); Gansu provincial hospital of TCM (Unknown); Tibet Autonomous Region People's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: ZS-3560
Record Dates: First submitted 2022-07-24; First posted 2022-07-26 (Actual); Last update posted 2024-05-13 (Actual); Status verified 2024-05

CONDITIONS: Pain, Postoperative
Keywords: Video-assisted thoracic surgery; Chronic post-surgical pain; Epidemiology study; risk factors
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is a nationwide multi-center study to investigate the incidence and risk factors of chronic post-surgical pain (CPSP) after receiving video-assisted thoracic surgery (VATS). Patients receiving VATS in participating centers across China in Aug. 2022 will be assessed for eligibility, and all the enrolled patients will be followed up for at least 6 months. The study's primary outcome is the incidence of CPSP 6 months after VATS. Baseline demographic, psychological , surgical, anesthesia-related and pain-related characteristics will be evaluated for possible risk factors of CPSP after VATS.

DETAILED DESCRIPTION:
Study Overview This is a multi-center perspective cohort study on the incidence and risk factors of CPSP after VATS.

Study aims

1. Investigate the incidence of chronic post-surgical pain in Chinese population who received video-assisted thoracic surgery by carrying out a multi-center, perspective cohort study
2. Perform regression analysis to evaluate the risk factors for chronic post-surgical pain in video-assisted thoracoscopic surgery.
3. Establish a risk-prediction model for CPSP after VATS

Time frame:

We plan to recruit patients from Aug 1st, 2022 to Sept 1st, 2022. And our follow-up will be performed at 1 month, 3 months and 6 months after the surgeries. After completing the follow-up of all patients, we are going to build a risk-prediction model and have it validated.

Study subjects Our research focuses on the incidence of CPSP after VATS in Chinese population. To select an accessible population that can well represent the target population, we set geographic criteria as regional medical centers in all seven geographical subregions of China, namely northwestern China, northern China, northeastern China, central China, southern China, southwestern China and southeastern China. Considering the needed sample size and the cost, we set time criteria as one month.

Plan for sampling As described before, our study plans to sample all the patients receiving VATS in participating medical centers across China for one month.

Plan for recruitment All patients receiving VATS in our participating centers will be examined for recruitment by the local coordinators according to our inclusion and exclusion criteria.

Plan for retaining subjects We are going to follow up the patients for at least 6 months after the surgery. At the pre-Op visit, the patient will be informed of the study time frame and he/she will be called by researcher in PUMCH during their follow-up. After their discharge, we will contact the patients and call them at 1, 3, 6 months after surgery.

Patient Registries We will use standard case report form (CRF) and electronic data capture (EDC) system for patient registries. All the data required in this study will be obtained by patient interview and medical records and recorded in our CRF and uploaded into EDC system. Researchers in participating centers will collect patient information by interview during their stay at the hospital. An SOP and interviewer training session will be developed for the study. The EDC system will help with data check, data dictionary. And our data monitoring board in PUMCH will check the uploaded data while follow-up telephoning the patients.

Statistical analysis plan Sample size Expected incidence: 30% Comment: the average reported incidence of CPSP after VATS Desired precision: 10% (total width) Confidence level: 95% Therefore, the estimated sample size with the above-mentioned parameters is 323 The risk factors will be analyzed by Logistics regression.

ELIGIBILITY:
Inclusion Criteria:

* In-patients at participating medical centers
* Scheduled for unilateral VATS during the study enrollment period

Exclusion Criteria:

* Emergency surgeries
* Patients with known pain sensory impairment
* Patients cannot express themselves so that an NRS score cannot be measured

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Our research focuses on the incidence of CPSP after VATS in Chinese population. So, our target population will be all the Chinese patients receiving VATS in China. To select an accessible population that can well represent the target population, we set geographic criteria as regional medical centers in all seven geographical subregions of China, namely northwestern China, northern China, northeastern China, central China, southern China, southwestern China and southeastern China. Considering the needed sample size and the cost, we set time criteria as one month.
  Therefore, the accessible population in our study is all the patients receiving VATS in Aug., 2022 at selected medical centers in all seven geographical subregions of China.
Sampling Method: Non-Probability Sample
Enrollment: 886 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
post-surgical pain-6 month | 6 month after the VATS
  Asking patients about the existence of chronic pain related to surgery by telephone interview

SECONDARY OUTCOMES:
post-surgical pain-3 month | 3 month after the VATS
  Asking patients about the existence of chronic pain related to surgery by telephone interview
Influence on quality of life | 3\6 month after the VATS
  Assessed by BPI-SF influence part

CONTACTS AND LOCATIONS:
Overall Officials: Le Shen, M.D., Ph.D., Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
In terms to patient's privacy, only the overall statistics will be reported. (i.e. incidence, risk factors, demographic characteristics). Individual date will not be available to other researchers.